CLINICAL TRIAL: NCT04819074
Title: The Prediction of Adverse Events After Microsurgery for Intracranial Unruptured Aneurysms (PRAEMIUM) Study
Brief Title: Prediction of Outcomes After Surgery for Unruptured Intracranial Aneurysms
Acronym: PRAEMIUM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: Macquarie University, Australia (Other); University of Melbourne (Other); Kepler University Hospital (Other); Medical University Innsbruck (Other); General University Hospital, Prague (Other); Universitätsklinikum Köln (Other); Goethe University (Other); University Medical Center Mainz (Other); University of Göttingen (Other); University Hospital Dresden (Other); Charite University, Berlin, Germany (Other); Heinrich-Heine University, Duesseldorf (Other); University of Roma La Sapienza (Other); University of Padova (Other); University of Florence (Other); Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other); University of Messina (Other); Universita di Verona (Other); University of Genua, Italy (Other); Leiden University Medical Center (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); UMC Utrecht (Other); Burdenko Neurosurgery Institute (Other); Sahlgrenska University Hospital (Other); University of Bern (Other); Barrow Neurological Institute (Other); Stanford University (Other); Emory University (Other); University of Wisconsin, Madison (Other); University of California, San Francisco (Other); University of Illinois at Chicago (Other); Brigham and Women's Hospital (Other); Mayo Clinic (Other); University of California, Los Angeles (Other); Endeavor Health (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: PRAEMIUM
Record Dates: First submitted 2021-03-18; First posted 2021-03-26 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Aneurysm, Brain
Keywords: machine learning; unruptured aneurysm
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Microsurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with unruptured brain aneurysms: We will include all adult patients (18 years or older) undergoing microsurgical treatment for UIAs. No specific exclusion criteria will be set. Patients with prior SAH may only be included when surgical treatment occurred at least 4 weeks after ictus. Only patients treated from January 1st 2010 onwards can be included in this study.
  No intervention.
  Interventions: Procedure: Microsurgery

INTERVENTIONS:
Procedure: Microsurgery — Microsurgery for unruptured intracranial aneurysm

SUMMARY:
Accurate preoperative identification of patients at high risk for adverse outcomes would be clinically advantageous, as it would allow enhanced resource preparation, better surgical decision-making, enhanced patient education and informed consent, and potentially even modification of certain modifiable risk factors. The aim of the Prediction of adverse events after microsurgery for intracranial unruptured aneurysms (PRAEMIUM) study is therefore to develop and externally validate a clinically applicable, robust ML-based prediction tool based on multicenter data from a range of international centers.

DETAILED DESCRIPTION:
Introduction Unruptured intracranial aneurysms (UIAs) are incidentally detected at an increasing rate, mostly owing to the rise in availability of non-invasive cranial imaging. Decision-making in UIAs is complex and requires consideration of many risk factors for aneurysm growth and rupture to balance the benefits and risks of treatment versus observation. This is due to: 1) the high morbidity and case fatality inherent to aneurysmal subarachnoid hemorrhage (SAH) 2) the relatively low rupture rate of unruptured aneurysms; 3) the potential morbidity and mortality rate associated with either microsurgical or endovascular treatment.

Some consistent risk factors for rupture have been identified, including involvement of the posterior circulation, larger diameter, higher age, and some specific populations such as Japanese and Finnish patients. Many other risk factors have been suggested based on varying levels of evidence. However, it is difficult to integrate this considerable number of factors into a single risk assessment and to present a clear clinical decision making algorithm to patients. A range of scoring systems have been developed and validated to approximate the risk of rupture (PHASES) and growth (ELAPSS) or to balance the risks and benefits of microsurgical treatment versus follow-up imaging directly (UIATS) by integrating some of these risk factors. Still, these scores are focused on predicting rupture events instead of neurological outcome. In addition, they usually are focused on solely one outcome, instead of providing a wide range of objective predictive analytics that may then improve shared decision-making.

Machine learning (ML) methods have been extraordinarily effective at integrating many clinical patient variables into one holistic risk prediction tailored to each patient. A previous pilot study has been carried out to assess the feasibility of predicting surgical outcomes after surgery for UIAs in a small single-center sample, and it was found that prediction was feasible with good performance metrics, and the most important factors to be included in such models were also identified. A robust, multicenter, externally validated prediction model or predictive score for surgical outcome after microsurgery for UIAs does not yet exist.

Methods Data will be collected by a range of international centers. Overall, the model will be built and publication will be compiled according to the transparent reporting of a multivariable prediction model for individual prognosis or diagnosis (TRIPOD) guidelines.

Each center will collect their data either retrospectively, or from a prospective registry, or from a prospective registry supplemented by retrospectively collected variables. Data from patients operated from January 1st 2010 and onwards will be eligible for inclusion. Data collection should be completed, and deidentified data should be sent to the sponsor institution.

A standardized Excel spreadsheet will be provided by the sponsor. The data will be entered in standardized and anonymized form. This spreadsheet will only contain a study-specific patient number. The data set is anonymized source data that includes clinical data extracted from electronic health records (retrospectively or from a prospective registry of already existing data). The data will be anonymized upon entering them into the PRAEMIUM Excel spreadsheet, after which the patients will be numbered consecutively and there will be no way to trace the data back to individual patients. No identifiable data such as date of birth will be included. Whenever the PRAEMIUM Excel spreadsheet is transferred, it will be encrypted using a password and sent through a secure institutional e-mail server. The password will be sent in a separate e-mail. Some missing data is acceptable, but should be kept to a minimum (i.e. must be < 10%)

Endpoint Definitions Models will be developed for the following three endpoints at discharge: Poor neurological outcome (1), as well as presence of (2) new sensorimotor neurological deficits and (3) any complications (surgical or non-surgical). Neurological outcome was assessed by the modified Rankin scale (mRS), and a favorable neurological outcome was defined as mRS 0, 1, or 2. Complications will be assessed using the modified 2009 Clavien-Dindo grading (CDG), and occurrence of a complication was defined as any deviation from CDG 0.The Clavien-Dindo grading system is a classification of surgical complications: Grad 0 signifying no complication, Grade I identifying complications with any deviation from the normal intra- or postoperative course requiring medical treatment, and so forth. Detailed definitions are provided in the Excel spreadsheet. Surgery-related as well as none-surgery-related complications are counted. In case of multiple complications, only the complication with the highest CDG was counted per patient.

Input Feature Definitions All features are measured preoperatively. Recorded baseline variables will include age, gender, maximum aneurysm diameter, anatomical location (artery), total number of aneurysms per patient, if multiple aneurysms were treated during the index session, calcification of the aneurysm wall or neck, aneurysm morphology (saccular, dissecting, fusiform, or other), involvement of critical perforating or branch vessels, and intraluminal thrombosis.

In addition, the investigators will capture prior SAH, mRS at admission, prior aneurysm treatment, presence of anticoagulation/antiplatelet therapy preoperatively, and hypertension, as well as American Society of Anesthesiologists (ASA) grading, the PHASES, ELAPSS, and UIATS scores including the UIATS "pro-repair" and "pro-conservative treatment" subscores. The unruptured intracranial aneurysm treatment score (UIATS) consists of two subscores: One that represents the strength of recommendation for invasive repair of an unruptured aneurysm, and one that represents the strength of recommendation for conservative management of an unruptured aneurysm. The final overall UIATS score is subsequently calculated as the difference between the two subscores. Also included was the surgical approach: minimally invasive or standard approach, and whether a bypass was performed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 or older)
* Undergone microsurgical treatment for unruptured intracranial aneurysm
* Patients with prior SAH may only be included when surgical treatment occurred at least 4 weeks after ictus.
* Treated from January 1st 2010 onwards

Exclusion Criteria:

* No specific exclusion criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We will include all adult patients (18 years or older) undergoing microsurgical treatment for UIAs. No specific exclusion criteria will be set. Patients with prior SAH may only be included when surgical treatment occurred at least 4 weeks after ictus. Only patients treated from January 1st 2010 onwards can be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale | Within 24 hours of admission to discharge, assessed up to 30 days
  Neurological outcome was assessed by the modified Rankin scale (mRS), and a favorable neurological outcome was defined as mRS 0, 1, or 2. The scale runs from 0 to 5, and higher scores mean a worse outcome.
Sensorimotor neurological deficits | Within 24 hours of admission to discharge, assessed up to 30 days
  Any new sensorimotor neurological deficits after surgery will be captured.
Clavien Dindo Complication Grading | Within 24 hours of admission to discharge, assessed up to 30 days
  Complications will be assessed using the modified 2009 Clavien-Dindo grading (CDG), and occurrence of a complication was defined as any deviation from CDG 0. The CDG runs from 0 to 5, and higher scores mean a worse complication.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Staartjes, Principal Investigator — USZ; Giuseppe Esposito, Principal Investigator — USZ
Locations (37):
- United States (10):
  - Barrow Neurological Institute, Phoenix, Arizona
  - UCLA, Los Angeles, California
  - UCSF, San Francisco, California
  - Stanford University, Stanford, California
  - Emory University Hospital, Atlanta, Georgia
  - University of Illinois, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - North Shore University Hospital, Manhasset, New York
  - University of Wisconsin, Madison, Wisconsin
- Australia (2):
  - Royal Melbourne Hospital, Melbourne
  - Macquarie University, Sydney
- Austria (2):
  - Innsbruck University, Innsbruck
  - Linz Kepler Klinikum, Linz
- Prague University, Prague, Czechia
- Germany (7):
  - Charité Univesitätsmedizin, Berlin
  - University of Cologne, Cologne
  - Dresden Uniklinikum, Dresden
  - Düsseldorf Universitätsmedizin, Düsseldorf
  - Frankfurt University, Frankfurt
  - Universitätsmedizin Göttingen, Göttingen
  - Unimedizin Mainz, Mainz
- Italy (8):
  - University of Florence - Careggi, Florence
  - University of Genoa, Genoa
  - University of Messina, Messina
  - Carlo Besta, Milan
  - Padova University, Padua
  - Gemelli University Hospital, Roma
  - Sapienza University, Roma
  - University of Verona, Verona
- Netherlands (3):
  - Amsterdam UMC, Amsterdam
  - Leiden University, Leiden
  - UMC Utrecht, Utrecht
- Burdenko Hospital, Moscow, Russia
- Sahlgrenska Hospital, Gothenburg, Sweden
- Switzerland (2):
  - Inselspital Bern, Bern
  - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT04819074/Prot_SAP_000.pdf